CLINICAL TRIAL: NCT00930566
Title: Allogenic Hematopoietic Stem Cell Transplantation (HSCT) From a Genoidentical Donor After a Reduced Intensity Conditioning Transplantation (RICT) Followed by an Early Preventive Treatment (Day 21) With Extracorporal Photopheresis After Transplantation.
Brief Title: Extracorporal Photopheresis Pilot Study
Acronym: ECP
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2006.409
Record Dates: First submitted 2009-06-29; First posted 2009-06-30 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2013-04

CONDITIONS: Hematological Malignancies
Keywords: Allogeneic Hematopoietic Stem Cell Transplantation; Extracorporeal Photopheresis
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Methoxsalen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Extracorporal Photopheresis (Experimental)
  Interventions: Drug: methoxsalen; Procedure: Extracoporal Photopheresis (ECP)

INTERVENTIONS:
Drug: methoxsalen — UVADEX® is supplied in a 10 mL single-use vial. Each mL of solution contains 20 mcg of UVADEX®.
  In the ECP process, UVADEX® will be injected directly into the Recirculation Bag of the extracorporal circuit after completion of the buffy coat collection, just prior to pressing the photoactivation button. The dose of UVADEX used to inoculate these cells will be calculated based on the treatment volume collected during the plasma/buffy coat collection process, usinge the following formula :
  Treatment Volume in mL x 0.017 = Dose of UVADEX® (in mLs) required for administration into the recirculation bag.
  After the cells are inoculated with UVADEX, the buffy coat/plasma suspension is irradiated with ultraviolet-A light and then reinfused back into the patient.
  Other Names: UVADEX®
Procedure: Extracoporal Photopheresis (ECP) — In the ECP process, UVADEX® will be injected directly into the Recirculation Bag of the extracorporeal circuit after completion of the buffy coat collection, just prior to pressing the photoactivation button.
  After the cells are inoculated with UVADEX, the buffy coat/plasma suspension is irradiated with ultraviolet-A light and then reinfused back into the patient.
  Other Names: ECP kits : UVAR®XTS™

SUMMARY:
ECP will be given to the patients [UVAR®XTS TM Therakos system, Johnson & Johnson] according to the following schedule:

Starting at day 21 after transplant, if hematologic recovery allowed it: 2 ECP per week the first 2 weeks, and 1 ECP per week during 1 month.

Total = 8 ECP after transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years and < or = 65 years with an hematological malignancy indicated for an allogeneic transplantation after reduced intensity conditioning :
* due to the age : for patients between 55 and 65 years.
* or for patients between 18 and 55 years of age presenting a risk of increased toxicity for myeloablative conditioning (cardiac, renal or pulmonary pathology)
* CML and MPS in blastic phase achieving CR,
* MM stage II or III, relapse after autologous transplant, achieving a response ≥ 30% or on first line if high risk,
* NHL in 2nd CR, PR after chemotherapy or autologous transplant, chemo-sensible.
* CLL in 2nd CR, PR after chemotherapy or autologous transplant, chemo-sensible.
* AML in 2nd CR or in first line for high risk criteria, secondary AML. In AML, high risk criteria are defined by : LAM 7, leukocytes>30000/mm3, cytogenetic abnormalities: t(6,9); 11q23, 17p, 11q, 20q, 21q, -5, del(5q), -7/del7q, del 9q and inv 3q,
* ALL in 2nd CR or in first line for high risk criteria defined by cytogenetic abnormalities: 11q23, t(9,22); t(1,19); t(4,11).
* MDS patients without prior chemotherapy
* HLA identical sibling donor
* Performans status < or = 2
* Patients member of a social security company

Exclusion Criteria:

* Age < 18 years or > 65 years
* Pregnant or lactating females
* Known HIV positivity
* Active infectious hepatitis, type A, B or C
* Performance status > 2 according to WHO
* Left ventricular ejection fraction < 40% and Alveolus-capillary diffusion < 50%
* Uncontrollable hypertension with medical therapy
* Creatinine clearance < 60 ml/min
* Hypersensitivity or allergy to psoralen (methoxsalen)
* Disease associated with a photosensitivity
* Hypersensitivity or allergy to both heparin and citrate products
* Contra-indication to Busulfan, Fludarabine, SAT or methotrexate
* Hypersensitivity to ciclosporine, mycophenolate mofetil or mycophenolic acid

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-04; Primary Completion 2011-09 (Actual); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the toxicity at Day 100 (NCI/NIH Common Toxicity Criteria) of Extracorporal Photopheresis (ECP) administered for Graft-versus-host-disease (GVHD) prophylaxis and introduced early (Day 21) after an HSCT from a genoidentical donor. | Day 100
  All types of toxicity will be assessed and graded according to NCI/NIH Common Toxicity Criteria

SECONDARY OUTCOMES:
Efficacy: decrease in incidence of acute GVHD and chronic GVHD | during 2 years
Incidence of Infection (clinically et/or bacteriologically proved) | during 2 years
Documentation of chimerism [quantification of donor-type chimerism in bone marrow and/ or in peripheral blood (total blood, CD3+)] | during 2 years
Transplant-related Mortality | at 3 months and 1 year
  TRM at 3 months for acute GVHD and at 1 year for chronic GVHD
Toxicity at Day 180 after HSC transplantation | Day 180
Disease-free survival (DFS) | at 1 and 2 years
progression-free survival (PFS) | at 1 and 2 years
Overall survival (OS) | at 1 and 2 years
cumulative incidence of relapse | at 1 and 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Mauricette Michallet, Professor, Principal Investigator — Hospices Civils de Lyon; Olivier Hequet, MD, Principal Investigator — Etablissement Français du Sang
Locations (2):
- France (2):
  - Centre de Santé - Etablissement Français du Sang (EFS), Lyon
  - Hôpital Edouard Herriot, Service d'Hématologie, Lyon